CLINICAL TRIAL: NCT06918067
Title: Comparison of Urinary Flow Speed Using 14 Fr Two Eyelet Coloplast Female SpeediCath Urinary Catheter Versus 14 Fr Coloplast Micro Zone Luja Female Catheter in Female Patients Using Intermittent Catheters
Brief Title: Comparison of Urinary Flow Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00128923
Record Dates: First submitted 2025-04-03; First posted 2025-04-09 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-03

CONDITIONS: Urinary Retention
Keywords: catheter; intermittent catheterization; bladder
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Luja / SpeediCath (Active Comparator): Subjects randomized to this arm will perform intermittent self-catheterization using the Coloplast Micro Zone Luja Female Catheter first then have bladder backfilled with sterile fluid to the amount equal to the volume of first catheterization. Then the subject will perform intermittent self-catheterization using the Coloplast Female SpeediCath Urinary Catheter.
  Interventions: Device: Coloplast Micro Zone Luja Female Catheter; Device: Coloplast SpeediCath Female Catheter
- SpeediCath / Luja (Active Comparator): Subject randomized to this arm will perform intermittent self-catheterization using the Coloplast Female SpeediCath Urinary Catheter first then have bladder backfilled with sterile fluid to the amount equal to the volume of first catheterization. Then the subject will perform intermittent self-catheterization using the Coloplast Micro Zone Luja Female Catheter.
  Interventions: Device: Coloplast Micro Zone Luja Female Catheter; Device: Coloplast SpeediCath Female Catheter

INTERVENTIONS:
Device: Coloplast Micro Zone Luja Female Catheter — clean self-catheterization with 14 Fr Coloplast micro zone Luja female urinary catheter
Device: Coloplast SpeediCath Female Catheter — clean self-catheterization with 14 Fr two eyelet Coloplast SpeediCath female urinary catheter

SUMMARY:
The purpose of this research study is to compare the urinary flow speed of two different female catheters in patients that use intermittent catheters to empty their bladder. The "14 Fr Two Eyelet Coloplast Female SpeediCath Urinary Catheter" will be compared to the "14 Fr Coloplast Micro Zone Luja Female Catheter." Participants will have one study visit that should take about an hour and will also receive a follow-up telephone call about one week after the visit.

DETAILED DESCRIPTION:
The purpose of this crossover study is to compare the urinary flow speed of two different female catheters manufactured by Coloplast, the "14 Fr Two Eyelet Coloplast Female SpeediCath Urinary Catheter" vs "14 Fr Coloplast Micro Zone Luja Female Catheter" in patients that use intermittent catheters to empty their bladder. Patients will be randomly assigned to group A or group B using a closed-envelope randomization method. Group A will self catheter with Luja, backfill with sterile fluid volume equal to amount of urine collected, then self-catheter with SpeediCath. Group B will self catheter with SpeediCath, backfill with sterile fluid volume equal to amount of urine collected, then self-catheter with Luja. Outcomes will be measured with office uroflow device.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Regular use of intermittent catheters to empty bladder, for at least 1 month before enrolment
* Age 18 years or older
* Required to adhere to the intervention procedure and not participate in any other clinical studies throughout the duration of this study

Exclusion Criteria:

* Severe urinary tract abnormalities (e.g. excessive production of urinary mucus/sediments/debris)
* Hypersensitive to the ingredients in the catheters being tested
* Recent surgery, within 3 months
* Currently being treated for urinary tract infection
* Being pregnant or breastfeeding
* Non-English speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — biologic females
Enrollment: 17 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Urinary flow duration | Day 1
  Amount of time (seconds) it takes the urine to be released. The normal urinary flow duration for women is 15-18 ml/sec. A lower average flow rate could indicate a problem with the bladder or urinary tract.
Total Urine Volume | Day 1
  total urine volume (mL) measured by uroflow device
Peak Flow Rate | Day 1
  Peak flow (mL/sec) measured by uroflow device. Normal peak urine flow rates typically range from 15 to 25 mL/sec for women. Reduced flow rates or a slow stream can indicate urinary tract obstruction or other issues.
Time to Peak Flow | Day 1
  Time (seconds) to peak flow measured by uroflow device. A normal peak flow rate for women is typically between 15 and 25 mL/sec. A lower rate may indicate a blockage or obstruction in the urinary tract.
Mean Flow | Day 1
  Mean flow (mL/sec) measured by uroflow device. Normal mean urine flow rates typically range from 15 to 25 mL/sec for women. A slow or low flow rate may mean there is an obstruction at the bladder neck or in the urethra or a weak bladder.
Total Urine voiding time | Day 1
  Total time (seconds) to void urine from beginning of urine flow to the end of flow, measured by uroflow device.

SECONDARY OUTCOMES:
Measuring patient's satisfaction of using catheter-Part a | Day 1
  Patient's preference of catheter type by using the Patient Global Impression of Improvement (PGI-I) scale
Measuring patient's satisfaction of using catheter-Part b | Day 1
  Patient's Satisfaction and Comments on Use of Luja Catheter

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kennelly, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Women's Center for Pelvic Health (Mercy), Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No